CLINICAL TRIAL: NCT03266848
Title: Quantitative Non-Invasive Brain Imaging Using QUTE-CE MRI
Status: Completed | Type: Observational
Sponsor: Theranano LLC (Industry)
Collaborators: Massachusetts General Hospital (Other); Northeastern University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: R41DA043974 (NIH); R41DA043974 (NIH)
Record Dates: First submitted 2017-08-16; First posted 2017-08-30 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Cerebrovascular Disorders
Keywords: Magnetic Resonance Imaging; Ferumoxytol
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subject blood sample before each scan
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Quantitative Magnetic Resonance Imaging — Radiological diagnosis

SUMMARY:
This trial will evaluate a non-invasive brain imaging technique QUTE-CE MRI and validate the method with first-in-human studies.

DETAILED DESCRIPTION:
This trial will evaluate a non-invasive brain imaging technique QUTE-CE MRI using Ferumoxytol as a contrast agent, and validate the method with first-in-human studies. Subjects who are already scheduled to receive ferumoxytol infusion will undergo MRI scans after the infusion. The ferumoxytol infusion itself is not a part of the study. The project will provide brain angiograms and establish a human cerebrovascular atlas that will enable future quantitative diagnosis of cerebrovascular abnormalities by revealing abnormal regions of the brain that characterize disease, a tool which doesn't currently exist, and which could lead to many exciting discoveries and clinical applications in neurology.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 to 80;
* Able to understand written consent document and HIPAA authorization prior to initiation of study related procedures.

Exclusion Criteria:

* Known allergy to ferumoxytol or any intravenous iron preparation;
* Iron saturation above the upper limit of normal;
* Individuals with a contraindication to MRI, such as the presence of metallic prostheses or implanted metal device (e.g., infusion pump, defibrillator);
* Individuals with known clinical conditions that may lead to iron overload including hemochromatosis, cirrhosis, or sickle cell disease;
* Individuals with any serious medical condition that the investigator believes may place them at increased risk for an adverse event.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with iron deficiency anemia already scheduled to receive ferumoxytol infusion for iron replacement therapy.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Cerebrovascular Angiography | 0-4 hours after ferumoxytol infusion
  Obtain angiograms of the cerebral vasculature from the MRI intensity data

SECONDARY OUTCOMES:
Quantitative cerebral blood volume atlas | 0-4 hours after ferumoxytol infusion
  Create cerebral blood volume atlas from the quantitative MRI intensity data

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Sridhar, Ph.D., Principal Investigator — Theranano LLC
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Timms L, Zhou T, Qiao J, Gharagouzloo C, Mishra V, Lahoud RM, Chen JW, Harisinghani M, Sridhar S. Super High Contrast USPIO-Enhanced Cerebrovascular Angiography Using Ultrashort Time-to-Echo MRI. Int J Biomed Imaging. 2024 Apr 13;2024:9763364. doi: 10.1155/2024/9763364. eCollection 2024. PMID 38644981